CLINICAL TRIAL: NCT01004315
Title: A Randomized, Double Blind, Placebo Controlled, Phase III Study of KUC-7483 in Patients With Overactive Bladder
Brief Title: A Confirmatory Study of KUC-7483 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUC1301
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Frequency; Micturition; Urgency; Urge urinary incontinence; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — ritobegron ethyl; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KUC-7483 (Experimental)
  Interventions: Drug: KUC-7483
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tolterodine (Active Comparator)
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: KUC-7483
  Arms: KUC-7483
Drug: Placebo
  Arms: Placebo
Drug: Tolterodine
  Arms: Tolterodine

SUMMARY:
To evaluate the efficacy and the safety of KUC-7483 in overactive bladder patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptom of overactive bladder for more than 6 months.
* Patients who meet the following condition during the 3-day bladder diary period.

  * the mean number of micturitions per 24 hours is ≥8 times
  * the mean number of urgency episodes per 24 hours is ≥1 time

Exclusion Criteria:

* Patients who are diagnosed as stress urinary incontinence are predominant.
* Patients with urinary calculus, interstitial cystitis, or clinically significant urinary tract infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean number of micturitions per 24 hours | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in the mean number of urgency episodes per 24 hours | 12 weeks
Change from baseline in the mean number of incontinence episodes per 24 hours | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Omori, Study Director — Clinical Development Department, Kissei pharmaceutical Co., Ltd.
Locations (1):
- Japan, Hokkaido,Tohoku,Kanto,Chubu,Kansai,Shikoku,Kyushu, Japan